CLINICAL TRIAL: NCT03112577
Title: A Randomized, Placebo-controlled, Parallel Panel Study to Assess the Effects of REGN3500, Dupilumab, and Combination of REGN3500 Plus Dupilumab on Markers of Inflammation After Bronchial Allergen Challenge in Patients With Allergic Asthma
Brief Title: Study of REGN3500 and Dupilumab in Patients With Asthma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R3500-AS-1633; 2016-003165-26 (EudraCT Number); SAR440340 (Other: Sanofi)
Record Dates: First submitted 2017-04-04; First posted 2017-04-13 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Asthma, Allergic
MeSH Terms: conditions — Asthma | interventions — itepekimab; dupilumab; Fluticasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- REGN3500 (Experimental): REGN3500: masked and randomized dosing regimen per protocol (part 1 only)
  Interventions: Drug: REGN3500
- Dupilumab (Experimental): Dupilumab: masked and randomized dosing regimen per protocol (part 1 only)
  Interventions: Drug: Dupilumab
- REGN3500 plus dupilumab (Experimental): REGN3500 plus dupilumab: masked and randomized dosing regimen per protocol (part 1 only)
  Interventions: Drug: REGN3500; Drug: Dupilumab
- Placebo (Experimental): Placebo: masked and randomized dosing regimen per protocol (part 1 only)
  Interventions: Drug: Placebo
- Fluticasone propionate (Active Comparator): Fluticasone propionate: open label dosing regimen per protocol (part 2 only)
  Interventions: Drug: Fluticasone propionate

INTERVENTIONS:
Drug: REGN3500 — Intravenous (IV) use
  Arms: REGN3500; REGN3500 plus dupilumab
Drug: Dupilumab — Subcutaneous (SC) use
  Other Names: Dupixent
  Arms: Dupilumab; REGN3500 plus dupilumab
Drug: Placebo — Matching placebo
  Arms: Placebo
Drug: Fluticasone propionate — Inhalation use
  Arms: Fluticasone propionate

SUMMARY:
To assess the effects of REGN3500, dupilumab, and REGN3500 plus dupilumab, compared with placebo, on changes in inflammatory gene expression signatures in sputum induced after a bronchial allergen challenge (BAC) in adults with mild allergic asthma, at week 4 after treatment initiation compared with those at screening.

ELIGIBILITY:
KEY Inclusion Criteria:

1. Male or female aged between 18 and 60 years
2. Has a Body Mass Index {BMI) of 17 to 33 kg/m2 at pre-study screening
3. Has a history of mild allergic asthma for at least 6 months
4. Is a non-smoker or ex-smoker for at least 12 months

KEY Exclusion Criteria:

1. Has a history of life-threatening asthma
2. Has been hospitalized or has attended the emergency room for asthma in the 12 months prior to screening
3. Has a history of severe allergies or history of an anaphylactic reaction
4. Has a history of drug or alcohol abuse within a year prior to the screening visit

Note: other protocol defined inclusion/exclusion criteria apply

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2019-03-20 (Actual); Study Completion 2019-12-09 (Actual)

PRIMARY OUTCOMES:
Difference in bronchial allergen challenge (BAC)-induced changes in sputum inflammatory markers in individuals treated with REGN3500, dupilumab and the combination of REGN3500 plus dupilumab or placebo | Screening (pre-treatment) to week 4 after treatment initiation

SECONDARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events (TEAEs) | Baseline to week 42
Severity of TEAEs | Baseline to week 42
Serum concentration-time profile of REGN3500 | Baseline to week 42
  Assessed by maximum plasma concentration [Cmax]
Serum concentration-time profile of REGN3500: Tmax (time at Cmax) | Baseline to week 42
Serum concentration-time profile of REGN3500: AUClast (area under the curve to the last measurable concentration) | Baseline to week 42
Immunogenicity of REGN3500 and dupilumab | Baseline to week 42
  Assessed by measurement of anti-drug antibodies (ADAs)
Serum concentration of total IL-33 after single IV dose | Up to Week 42
Difference in the BAC-induced changes in sputum inflammatory mRNA signature in individual patients treated with fluticasone | Screening (pre-treatment) to day 4 after treatment initiation

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (5):
- WCCT Global, Cypress, California, United States
- United Kingdom (4):
  - Celerion, Belfast
  - Hammersmith Medicine Research, London
  - Respiratory Clinical Trials Ltd, London
  - The Medicines Evaluation Unit, Manchester